CLINICAL TRIAL: NCT06704672
Title: Clinical Study to Evaluate the Impact of the Accu-Chek SmartGuide CGM Solution on the Mean Change in Time in Range of 70 - 180 mg/dl Compared to SMBG
Brief Title: Clinical Study to Evaluate the Impact of the Accu-Chek SmartGuide CGM Solution on the Mean Change in Time in Range Compared With Self-Monitoring of Blood Glucose in Participants With Type 1 and Type 2 Diabetes Mellitus
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Collaborators: Roche Diabetes Care (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DC000129
Record Dates: First submitted 2024-11-22; First posted 2024-11-26 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Type 1 Diabetes Mellitus; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A: Accu-Chek SmartGuide CGM Solution (Experimental)
  Interventions: Device: Accu-Chek SmartGuide CGM Solution
- Group B: Self-Monitoring of Blood Glucose (SMBG) (Other)
  Interventions: Device: Accu-Chek SmartGuide Sensor and Blinded Apps; Device: SMBG Device

INTERVENTIONS:
Device: Accu-Chek SmartGuide CGM Solution — The Accu-Chek SmartGuide CGM solution is used for real-time continuous glucose monitoring (CGM) in the interstitial fluid. It consists of the Accu-Chek SmartGuide device and two smartphone applications (apps): the Accu-Chek SmartGuide app and the Accu-Chek SmartGuide Predict app. The Accu-Chek SmartGuide device contains a CGM sensor pre-assembled in a sensor applicator. It has connectivity to the smartphone that is running the Accu-Chek apps. The Accu-Chek SmartGuide app is the primary display of the real-time glucose values. The Accu-Chek SmartGuide Predict app is an information management tool that further visualizes and analyzes diabetes data from the Accu-Chek SmartGuide device.
  Arms: Group A: Accu-Chek SmartGuide CGM Solution
Device: Accu-Chek SmartGuide Sensor and Blinded Apps — The participants in the SMBG control group will wear a SmartGuide sensor with blinded SmartGuide apps intermittently, i.e., during the assessment periods. It is not possible to read out the glucose data from the blinded app, hence neither the SmartGuide app nor the SmartGuide Predict functionalities can be accessed by the participants in this group.
  Arms: Group B: Self-Monitoring of Blood Glucose (SMBG)
Device: SMBG Device — With the SmartGuide apps in blinded mode, participants in the SMBG control group will continue using their own SMBG device or they may use the Accu-Chek Instant meter that will be provided for calibration of the SmartGuide device.
  Arms: Group B: Self-Monitoring of Blood Glucose (SMBG)

SUMMARY:
This is an open label, two-arm, randomized multi-center clinical device study in adult subjects with Type 1 diabetes (T1D) or insulin-dependent Type 2 diabetes (T2D) on a multiple daily injection (MDI) regime.

The goal of the study is to investigate the impact of the Accu-Chek SmartGuide CGM solution on the change in overall time in range (TIR) of blood glucose concentrations of 70-180 mg/dl compared with that using self-monitoring of blood glucose (SMBG).

ELIGIBILITY:
Inclusion Criteria:

* Type 1 Diabetes mellitus (T1D) or Type 2 Diabetes mellitus (T2D) diagnosed at least 12 months prior to screening, using multiple daily injection (MDI) regime for at least six months prior to screening
* Performing SMBG, no CGM/flash glucose monitoring (FGM) use during the last six months prior screening
* HbA1c ≥8% and ≤10% based on analysis from a local laboratory

Exclusion Criteria:

* Untreated adrenal or thyroid insufficiency
* Severe visual impairment
* Significant renal impairment: eGFR <30 ml/min within last one year
* Serious acute or chronic concomitant disease or an anamnesis which might, in the opinion of the investigator, pose a risk to the subject
* Hematocrit greater than 10% below the lower limit of normal
* Pregnancy (lack of negative pregnancy test - except in case of menopause, sterilization or hysterectomy - self-reported), planned pregnancy, or breast feeding
* Allergic to the adhesive (glue or tape)
* Skin diseases (e.g. psoriasis vulgaris, bacterial skin diseases) at the sensor application sites
* Sickle cell disease, or hemoglobinopathy
* Elective surgery planned that requires general anesthesia during study participation
* Current or anticipated acute uses of glucocorticoids (oral, injectable, or intravenous)
* Medical conditions that, per investigator determination, make it inappropriate or unsafe to target an HbA1c of <7%. Conditions may include but are not limited to: heart failure, unstable cardiovascular disease, recent myocardial infarction, ventricular rhythm disturbances, recent transient ischemic attack or cerebrovascular accident, significant malignancy
* Chronic use of opiates, opioids, morphinomimetics more than three times per week, which has not stopped at least 30 days prior to screening and any other medication interfering with the assessment of pain, as per investigator's discretion
* Intake of hydroxyurea (hydroxycarbamide), levodopa, methyldopa, ascorbic acid, acetylsalicylic acid (≥300mg), which has not stopped at least 30 days prior to screening
* Magnetic resonance tomography (MRT), computed tomography (CT), X-ray, radiofrequency ablation, high-frequency electrical heat or high intensity focused ultrasound planned during the course of the study
* Planned flight or high-altitude hike (>3000 m) during baseline and assessment periods
* Shift-worker (night-shifts)
* On or planning to start a diet intended for weight change
* Currently abusing illicit and/or prescription drugs or alcohol as judged by the investigator
* Any other physical or psychological disease or psychiatric disorder that could limit adherence to the required study tasks and interfere with the normal conduct of the study as judged by the investigator
* Dependency (e.g., employee, co-worker or family member) on sponsor, investigator or companies active in the field of CGM (e.g. Dexcom, Abbott, Menarini, Medtronic) or their subsidiaries
* Participation in another clinical study at the same time

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-06-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in the Percentage of Time in Range of a Blood Glucose Concentration of 70 to 180 mg/dL from the Baseline Period to Assessment Period A | Baseline Period (Weeks 1 and 2) and Assessment Period A (Weeks 5 and 6)

SECONDARY OUTCOMES:
Change in the Percentage of Time in Range of a Blood Glucose Concentration of 70 to 180 mg/dL from the Baseline Period to Assessment Period B | Baseline Period (Weeks 1 and 2) and Assessment Period B (Weeks 13 and 14)
Change in the Percentage of Time in Range of a Blood Glucose Concentration of 70 to 180 mg/dL from the Baseline Period to Assessment Period C | Baseline Period (Weeks 1 and 2) and Assessment Period C (Weeks 25 and 26)
Percentage of Time in Tight Range of a Blood Glucose Concentration of 70 to 140 mg/dL by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Percentage of Time Above Range (Blood Glucose Concentration of >180 to ≤250 mg/dL) in Level 1 Hyperglycemia by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Percentage of Time Above Range (Blood Glucose Concentration >250 mg/dL) in Level 2 Hyperglycemia by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Percentage of Time Below Range (Blood Glucose Concentration of ≥54 to <70 mg/dL) in Level 1 Hypoglycemia by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Percentage of Time Below Range (Blood Glucose Concentration <54 mg/dL) in Level 2 Hypoglycemia by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Number of Level 1 Hypoglycemia Events by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
  A level 1 hypoglycemia event is defined as a blood glucose concentration of ≥54 to <70 mg/dL for at least 15 minutes.
Number of Level 2 Hypoglycemia Events by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
  A level 2 hypoglycemia event is defined as a blood glucose concentration of <54 mg/dL for at least 15 minutes.
Average Glucose Management Indicator, as an Estimate of HbA1c, by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Average Blood Glucose Concentration by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Average Glycemic Variability in Blood Glucose Concentration by Study Period | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Average HbA1c Values from the Central Laboratory | Baseline (Week 1 Day 1), Week 15 Day 1, and Week 27 Day 1
Average Daily Insulin Dose | Baseline (Week 1), Weeks 5, 13, and 25
Average Number of Daily Insulin Boluses Injected | Baseline (Week 1), Weeks 5, 13, and 25
Average Daily Amount of Carbohydrates Consumed | Baseline (Week 1), Weeks 5, 13, and 25
Hypoglycemia Fear Survey-II (HFS-II) Score at Specified Timepoints | Baseline (Week 1 Day 1), Week 15 Day 1, and Week 27 Day 1
Diabetes Distress Scale 17 (DDS-17) Questionnaire Score at Specified Timepoints | Baseline (Week 1 Day 1), Week 15 Day 1, and Week 27 Day 1
Ecological Momentary Assessment (EMA) Questionnaire Score at Specified Timepoints | Baseline Period (Weeks 1 and 2), Assessment Periods A (Weeks 5 and 6), B (Weeks 13 and 14), and C (Weeks 25 and 26)
Number of Participants by Their Responses to the Roche Diabetes Care SmartGuide Usability Questionnaire (Group A Only) | Week 27 Day 1
Number of Healthcare Providers (HCP) by Their Responses to the Roche Diabetes Care HCP Accu-Chek Care Questionnaire | Week 27 Day 1

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (13):
- Poland (10):
  - Centrum Badań Klinicznych PI-House sp. z o.o., Gdansk
  - Diabetes Technology Center, Jagiellonian University Medical College, Krakow
  - NZOZ Neuromed, Kraśnik
  - NZOZ Neuromed, Lublin
  - Institute of Rural Health, Lublin
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - BioResearch Group Sp. z o. o., Nadarzyn
  - Nbr Polska, Warsaw
  - Clinic of Internal Diseases, Endocrinology and Diabetology State Medical Institute MSWiA, Warsaw
  - ETG Warszawa, Warsaw
- Turkey (Türkiye) (3):
  - Baskent University Department of Endocrinology and Metabolism, Adana
  - Bakırköy Sadi Konuk Training and Research Hospital, Bakirkoy Istanbul
  - Koç University Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: Yes
For eligible studies, qualified researchers may request access to individual patient level clinical data. See Roche's commitment to transparency of clinical study information here: https://go.roche.com/data_sharing